CLINICAL TRIAL: NCT03707626
Title: Does Coronary Collateral Circulation Mask the Presence of a Wellens Sign in Patients With Critical Stenosis of the Left Anterior Descending Artery?
Brief Title: Collateral Circulation to LAD and Wellens Sign
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Coney Island Hospital, Brooklyn, NY (Other)
Responsible Party: Principal Investigator, George Juang, Primary Investigator, Coney Island Hospital, Brooklyn, NY
Other Study IDs: 18-08-283-378(HHC)
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Coronary Artery Disease; Acute Myocardial Infarction; Acute Myocardial Infarction of Anterior Wall; Collateral Circulation, Any Site
Keywords: wellens sign; coronary collateral circulation; acute myocardial infarction; left anterior descending artery
MeSH Terms: conditions — Coronary Artery Disease; Anterior Wall Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LAD with collaterals with and without wellens sign
  Interventions: Other: Wellens Sign

INTERVENTIONS:
Other: Wellens Sign — presence or absence in presence of coronary collaterals to LAD

SUMMARY:
Overall Aim Coronary artery disease significantly contributes to morbidity and mortality in the United States. Atherosclerotic disease can lead to stenosis of the coronary arteries and subsequent cardiac hypoperfusion. Patients with a critical stenosis of the LAD, potentially leading to acute anterior wall myocardial infarction, may be asymptomatic at presentation with subtle EKG changes as its only manifestation. It is imperative for physicians to recognize patients with new T wave inversions in leads V2-V3 as the standard course of management may lead to poor prognosis.

The purpose of this study is to determine if collateral circulation to the left anterior descending (LAD) artery will mask the presence of a Wellens sign and therefore diminish its diagnostic utility. The conclusion of this study would raise awareness for physicians in light of an absent Wellens sign.

Hypothesis The presence of coronary collateral circulation to the LAD masks the presence of a Wellens sign (both Type 1 and Type 2) in precordial leads V2-V4.

DETAILED DESCRIPTION:
Introduction Electrocardiograms are an inexpensive and indispensible tool to assess cardiac rhythm and ischemia. A Wellens sign on an EKG is either a deeply inverted (Type 1) or biphasic (Type 2) t-wave in precordial leads V2-V3 (but may extend to other precordial leads). It is associated with critical stenosis of the proximal left anterior descending (LAD) artery. Patients with a Wellens sign are at high risk for extensive anterior wall myocardial infarction as the LAD is the main coronary artery that supplies the left ventricle. Exercise stress testing is contraindicated in this patient population. In addition, appropriate management of these patients is crucial to avoid acute myocardial infarction.

There have been a number of studies addressing the role of collateral coronary circulation in myocardial infarctions. Some studies show that the presence of collateral circulation is associated with improved in-hospital outcomes in patients following a ST-elevation myocardial infarction (STEMI) whereas others show that collateral circulation does not decrease morbidity and mortality in patients following acute STEMI. Similarly, patients with collateral circulation may have normal EKGs and be asymptomatic at rest but are symptomatic with corresponding abnormal EKG findings during periods of increased cardiac demand.

Patients with a critically stenosed LAD may be asymptomatic and have normal to minimally elevated cardiac enzymes at the time of presentation with at rest abnormal EKG findings being the sole clue to the patient's gravity. While some studies have shown collateral coronary circulation lead to normal EKGs, there is limited research addressing whether or not collateral circulation affects the presence of a Wellens sign. As a result, its diagnostic utility is questionable.

Overall Aim Coronary artery disease significantly contributes to morbidity and mortality in the United States. Atherosclerotic disease can lead to stenosis of the coronary arteries and subsequent cardiac hypoperfusion. Patients with a critical stenosis of the LAD, potentially leading to acute anterior wall myocardial infarction, may be asymptomatic at presentation with subtle EKG changes as its only manifestation. It is imperative for physicians to recognize patients with new T wave inversions in leads V2-V3 as the standard course of management may lead to poor prognosis.

The purpose of this study is to determine if collateral circulation to the left anterior descending (LAD) artery will mask the presence of a Wellens sign and therefore diminish its diagnostic utility. The conclusion of this study would raise awareness for physicians in light of an absent Wellens sign.

Study Objectives

To identify if coronary collateral circulation masks the presence of a Wellens sign by:

Evaluating catheterization reports Examining for the presence of coronary collateral circulation Examining EKGs for presence of deeply inverted t-waves in precordial leads Examining EKGs for presence of biphasic t-waves in precordial leads Correlating the presence/absence of coronary collateral circulation with EKG findings

Hypothesis:

The presence of coronary collateral circulation to the LAD masks the presence of a Wellens sign (both Type 1 and Type 2) in precordial leads V2-V4.

Study Design This study will be a retrospective chart review of patients who received cardiac catheterization and had LAD and/or Left Main lesions between the years 2000-2016 at Coney Island Hospital. Catheterization imaging and reports will be reviewed for collateral circulation. Subsequent pre-catheterization electrocardiograms, dated up to 1 year prior to cardiac catheterization, will be reviewed for the presence or absence of symmetrical deep (≥2 mV) t-wave inversion (type 1) or biphasic t-wave (type 2) Wellens sign in precordial leads. EKGs will be accessed either electronically or physically. All data will be de-identified and coded to maintain patient confidentiality.

What and how will you measure or collect data to test your hypothesis (or study objectives)? A retrospective chart review of cardiac catheterizations will be employed to assess the presence of coronary collateral circulation. Grading of coronary collateral circulation will be divided into four categories (0=no filling, 1=filling of side branches only, 2=partial filling of epicardial segments, 3=complete filling of epicardial segments). In addition, pre-catheterization EKGs will be analyzed for a.) the presence or absence of deeply inverted t-waves (type 1) or biphasic t-waves (type 2) and b.) the amplitude (mV) of each corresponding Wellens sign. Demographic data including medical record number, age, gender, and known risk factors, including but not limited to diabetes, smoking, drinking, previous myocardial infarction, hyperlipidemia, and hypertension, will be recorded for data analysis.

Describe where the research data will reside and who will have access to hold or maintain the data? Research data will be collected and recorded on a password protected Microsoft Excel Spreadsheet. Excel file will be saved on Coney Island Hospital servers. Computers are password protected and every effort will be made to ensure safekeeping of the aforementioned Excel file. File will be stored for a maximum of three years and will be permanantly eliminated following the conclusion and publication of proposed study.

Data will be managed by Dr. Ida Hui Suen and Dr. George Juang. Data will not be released to other collaborators. De-identified data will be forwarded to central office for assistance with statistical analysis if needed.

Describe the methods that will be used to destroy data and/or specimens at the end of the research study life cycle.

Efforts will be made to ensure that all files are deleted from Coney Island Servers. No specimens will be collected.

Data Analysis Statistical analysis will be performed with the assistance of Brian Altonen of New York Health and Hospital Corporation's Central Office. Chi Square, ANOVA, and multiple logistic regression analyses will be applied.

Sample Size Approximately 6,000 patients received cardiac catheterizations at Coney Island Hospital between 2003-2016. Approximately 30% will have LAD lesions (N=1800); of which approximately 20% will have a Wellens sign (N=360).

Variables Age, Nominal Sex, Categorical (1=M, 2=F) Date of Catheterization Location of Lesion, Categorical (1=LAD Proximal, 2=LAD Mid, 3=LAD Distal, 4=Left Main) Collaterals present, Categorical (0=N, 1=Y) Grading of Collaterals, Categorical (0=none, 1= filling of side branches, 2=partial filling of epicardial segment, 3=complete filling of epicardial segment) Date of pre-cath EKG Wellens Sign Present, Categorical (1=Y, 2=N) Type of Wellens Sign, Categorical (1=Type 1, 2=Type 2)

ELIGIBILITY:
Inclusion Criteria:

All patients receiving cardiac catheterization between 2003-2016 at Coney Island Hospital with LAD lesions and pre-catheterization electrocardiograms.

Exclusion Criteria:

None

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Coney Island Hospital between ages 18-89 years old between years of 2003-2016 receiving cardiac catheterization with pre-catheterization electrocardiograms
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-06-23 (Estimated); Study Completion 2019-06-23 (Estimated)

PRIMARY OUTCOMES:
Wellens Sign | 2003-2016

CONTACTS AND LOCATIONS:
Overall Officials: George Juang, MD, Principal Investigator — Coney Island Hospital
Locations (1):
- Coney Island Hospital, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Zwaan C, Bar FW, Wellens HJ. Characteristic electrocardiographic pattern indicating a critical stenosis high in left anterior descending coronary artery in patients admitted because of impending myocardial infarction. Am Heart J. 1982 Apr;103(4 Pt 2):730-6. doi: 10.1016/0002-8703(82)90480-x. PMID 6121481
- [Background] Haines DE, Raabe DS, Gundel WD, Wackers FJ. Anatomic and prognostic significance of new T-wave inversion in unstable angina. Am J Cardiol. 1983 Jul;52(1):14-8. doi: 10.1016/0002-9149(83)90061-9. PMID 6602539
- [Background] Yaylak B, Altintas B, Ede H, Baysal E, Akyuz S, Bilge O, Sevuk U, Erdogan G, Ciftci H. Impact of Coronary Collateral Circulation on In-Hospital Death in Patients with Inferior ST Elevation Myocardial Infarction. Cardiol Res Pract. 2015;2015:242686. doi: 10.1155/2015/242686. Epub 2015 Nov 25. PMID 26689135
- [Background] Gohlke H, Heim E, Roskamm H. Prognostic importance of collateral flow and residual coronary stenosis of the myocardial infarct artery after anterior wall Q-wave acute myocardial infarction. Am J Cardiol. 1991 Jun 1;67(15):1165-9. doi: 10.1016/0002-9149(91)90920-g. PMID 2035435
- [Background] Freedman SB, Dunn RF, Bernstein L, Morris J, Kelly DT. Influence of coronary collateral blood flow on the development of exertional ischemia and Q wave infarction in patients with severe single-vessel disease. Circulation. 1985 Apr;71(4):681-6. doi: 10.1161/01.cir.71.4.681. PMID 3971537
- [Background] Martinez-Rios MA, Da Costa BC, Cecena-Seldner FA, Gensini GG. Normal electrocardiogram in the presence of severe coronary artery sease. Am J Cardiol. 1970 Mar;25(3):320-4. doi: 10.1016/s0002-9149(70)80009-1. No abstract available. PMID 5443910